CLINICAL TRIAL: NCT00286871
Title: Steroid Avoidance in Hep C OLT
Brief Title: Randomized Controlled Trial in Liver Transplant Recipients Treated in Steroid Sparing Regimen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6538; 6538-04-11R0 (Other: Duke legacy protocol ID)
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2006-02

CONDITIONS: Chronic Hepatitis C; Organ Transplantation; Immunosuppression
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Cyclosporine; Tacrolimus

INTERVENTIONS:
Drug: Neoral
Drug: Tacrolimus

SUMMARY:
Liver transplant subjects will be given Mycophenolate (MMF) and Tacrolimus in order to help prevent post-transplant rejection.

DETAILED DESCRIPTION:
Recurrent HCV in the liver allograft is becoming the leading indicator for retransplantation. Studies suggest that glucocorticord-based immunosuppression regimens hasten the onset and progression of recurrent chronic HCV liver disease. Treatment of acute allograft rejection with steroid boluses is also associated with rapid HCV recurrence. The relative contribution of various calcineurin inhibitors to recurrent HCV liver disease has not been established. Previous retrospective studies, as well as prospective studies have not demonstrated a difference in recurrent HCV liver disease rates between patients receiving CsA or tacrolimus immunosuppression regimens respectively.

ELIGIBILITY:
Inclusion Criteria:

* adult patients who have received liver transplant

Exclusion Criteria:

* pregnant women
* nursing women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-02; Study Completion 2009-02

PRIMARY OUTCOMES:
compare timing & severity of recurrent chronic HCV disease Neoral versus Prograf

SECONDARY OUTCOMES:
compare the effectiveness of Neoral with Prograf as primary immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Devai Desai, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Gane EJ, Portmann BC, Naoumov NV, Smith HM, Underhill JA, Donaldson PT, Maertens G, Williams R. Long-term outcome of hepatitis C infection after liver transplantation. N Engl J Med. 1996 Mar 28;334(13):815-20. doi: 10.1056/NEJM199603283341302. PMID 8596547
- [Background] Berenguer M, Prieto M, Palau A, Rayon JM, Carrasco D, Juan FS, Lopez-Labrador FX, Moreno R, Mir J, Berenguer J. Severe recurrent hepatitis C after liver retransplantation for hepatitis C virus-related graft cirrhosis. Liver Transpl. 2003 Mar;9(3):228-35. doi: 10.1053/jlts.2003.50029. PMID 12619018
- [Background] McCaughan GW, Zekry A. Pathogenesis of hepatitis C virus recurrence in the liver allograft. Liver Transpl. 2002 Oct;8(10 Suppl 1):S7-S13. doi: 10.1053/jlts.2002.35856. PMID 12362292
- [Background] Zervos XA, Weppler D, Fragulidis GP, Torres MB, Nery JR, Khan MF, Pinna AD, Kato T, Miller J, Reddy KR, Tzakis AG. Comparison of tacrolimus with neoral as primary immunosuppression in hepatitis C patients after liver transplantation. Transplant Proc. 1998 Jun;30(4):1405-6. doi: 10.1016/s0041-1345(98)00291-7. No abstract available. PMID 9636568
- [Background] Eason JD, Loss GE, Blazek J, Nair S, Mason AL. Steroid-free liver transplantation using rabbit antithymocyte globulin induction: results of a prospective randomized trial. Liver Transpl. 2001 Aug;7(8):693-7. doi: 10.1053/jlts.2001.26353. PMID 11510013
- [Background] Knodell RG, Ishak KG, Black WC, Chen TS, Craig R, Kaplowitz N, Kiernan TW, Wollman J. Formulation and application of a numerical scoring system for assessing histological activity in asymptomatic chronic active hepatitis. Hepatology. 1981 Sep-Oct;1(5):431-5. doi: 10.1002/hep.1840010511. PMID 7308988